CLINICAL TRIAL: NCT00221689
Title: Early Treatment of Paroxysmal Dysautonomia and Hypertonia for Severe Brain Injured Patients by Intrathecal Baclofen Therapy
Brief Title: Intrathecal Baclofen Therapy and Paroxysmal Dysautonomia in Severe Brain-Injured Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: very slow recruitment and treatments beyond expiry date
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9244-01; 2001-009
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Traumatic Brain Injury; Cerebral Anoxia; Coma; Hypertonia; Dysautonomia
Keywords: Severe brain injury; Coma; Hypertonia; Dysautonomia; Baclofen; Randomized Controlled Trials
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypoxia, Brain; Coma; Muscle Hypertonia; Autonomic Nervous System Diseases; Brain Injuries | interventions — Baclofen; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: baclofen (drug)

SUMMARY:
Within the framework of a prospective double-blind and randomized study evaluating the efficacy of continuous intrathecal baclofen therapy (CIBT) on paroxysmal dysautonomia (main objective) and hypertonia, recovery and tolerance (secondary objectives) during the initial recovery phase of severe head injury, continuous intrathecal baclofen infusion will be delivered. The first week of study is double-blind: the first of two parallel groups receives CIBT and the second group receives placebo. The main outcome (number of neurovegetative episodes) is assessed at the end of first week. The second week of study is open labeled: active treatment is continued in the first group and the second group starts active CIBT treatment. The third week of study, treatment is stopped in both groups.

DETAILED DESCRIPTION:
Background. Severe brain trauma and especially serious brain lesions inducing coma lead to many cases of disability. A large number of these patients (about 30%) present neurovegetative and hypertonic episodes that are associated to a bad vital prognosis and the degree of disability. Several teams including two in France have reported the efficacy of intrathecal baclofen on such neurovegetative episodes that to date have not been able to be treated efficiently.

Objectives. The main objective of this trial is to assess the efficacy of infused intrathecal baclofen on the number of neurovegetative episodes in seriously brain-injured patients. The secondary aims are to evaluate the efficacy of the treatment on hypertonia, to assess changes in waking and treatment safety.

Study design. Double-blind randomized trial on two parallel groups. The second part of the study is open label: both groups receive the experimental treatment.

Intervention

Experimental group: continuous progressive dose of intrathecal baclofen for one week; constant dose of baclofen during the second week receives at a dose determined after the first week. Treatment is stopped after two weeks, but patients are assessed until the end of the third week.

Control group: intrathecal placebo for one week; progressive dose of intrathecal baclofen during the second week. Treatment is stopped after two weeks, but patients are assessed until the end of the third week.

Outcomes. The main outcome is the number of neurovegetative episodes in the last 48 hours of the first week of treatment. Secondary outcomes are hypertonia as measured by the Ashworth scale on D2 to D5 of all three weeks. Waking will be assessed by the WHIM scale on D5 each week. Adverse events are assessed throughout the 3 weeks of study.

Eligibility criteria. Inclusion criteria are focal or diffuse encephalic lesions leading to coma (Glasgow score <8), age 18 years or over, in waking phase (spontaneous eye-opening) since at least one month and less than six months, severe hypertonia of the lower members (mean Ashworth score >= 3) with neurovegetative episodes (at least 10 in 48 hours) and/or decortication after failure of treatment per os (clonidine, beta-blocker, baclofen per os). Non inclusion criteria are surgical, anesthetic or allergic contraindication to baclofen, uncontrolled sepsis directly threatening the implanted device or associated medullary trauma.

Expected results. Throughout the trial the patients will be hospitalized in the neurosurgical or neurological intensive care departments. Expected results are a very clear decrease in the number of neurovegetative episodes and a substantial reduction in hypertonia, at least in the lower limbs. It will also be possible to quantify the consequences of these improvements on waking.

ELIGIBILITY:
Inclusion Criteria:

* severe brain injury with coma (Glasgow score <8)
* Early phase of recovery (spontaneous eye-opening) since at least one month and less than six months
* severe hypertonia of the lower limbs (mean Ashworth score >= 3) with neurovegetative episodes (at least 10 in 48 hours) and/or decortication after failure of treatment per os (clonidine, beta-blocker, baclofen per os)
* written informed consent (next of kin)

Exclusion Criteria:

* surgical, anesthetic or allergic contraindication to baclofen
* uncontrolled sepsis directly threatening the implanted device
* associated medullary trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-03; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Number of neurovegetative episodes | day 6 and day 7

SECONDARY OUTCOMES:
Ashworth scale
Whim scale
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Cuny, Professor, Principal Investigator — University Hospital, Bordeaux; Paul Perez, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Service de neurochirurgie B, Hôpital Pellergin Tripode, Bordeaux, France